CLINICAL TRIAL: NCT06217159
Title: The Mechanistic Effect of Ketones on Cerebral Blood Flow and Cerebrovascular Function
Brief Title: Mechanistic Effect of Ketones on Cerebral Blood Flow
Acronym: MEKC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Jeremy Walsh, Assistant Professor, McMaster University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: MEKC
Record Dates: First submitted 2023-12-01; First posted 2024-01-22 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Cerebrovascular Function; Cerebral Blood Flow
Keywords: Cerebral Blood Flow; Beta-hydroxybutyrate (β-OHB); Cerebrovascular Function

STUDY DESIGN:
Intervention Model Description: A randomized single-blind crossover design will be used to test 2 conditions. Participants will consume 60 mL of a supplement containing 0.6g/kg body weight of the ketone monoester ([R]-3-hydroxybutyl [R]-3-hydroxybutyrate) in both conditions, and their PetCO2 will be maintained in the normocapnic conditions or not maintained in the poikilocapnic condition, in a randomized order.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Poikilocapnia (Sham Comparator): Room air-breathing
  Interventions: Dietary Supplement: Poikilocapnia
- Normocapnia (Experimental): Breathing air mixture with slightly elevated CO2 to maintain PetCO2 to resting baseline levels
  Interventions: Dietary Supplement: Normocapnia

INTERVENTIONS:
Dietary Supplement: Poikilocapnia — Following ingestion of 0.6 g β-OHB/kg body weight ketone monoester, participants will wear a specialized face mask and breathe room air for 60 min. The face mask will be attached to an automated gas-blender system; however, only room air will be delivered.
  Arms: Poikilocapnia
Dietary Supplement: Normocapnia — Following ingestion of 0.6 g β-OHB/kg body weight ketone monoester, participants will be outfitted with a specialized face mask and breathe air with a slightly higher concentration of CO2 to maintain PetCO2 to resting baseline values for 60 min. Gas will be continuously delivered by an automated gas-blender system.
  Arms: Normocapnia

SUMMARY:
Oral supplements containing exogenous ketones have recently become available and represent a novel tool for increasing plasma ketone bodies without the need for dietary restriction. Early evidence suggests that oral ketone supplements may enhance cerebral blood flow (CBF). However, a higher dose of a ketone monoester has been shown to slightly lower blood pH and reduce end-tidal CO2 (PetCO2) due to compensatory hyperventilation, which is accompanied by parallel reductions in CBF. Whether reductions in PetCO2 causes reductions in CBF is currently unknown.

The purpose of this study is to investigate the effect of manipulating PetCO2 at normocapnia (PetCO2 maintained at baseline) or poikilocapnia (no PetCO2 targeting; breathing room air), following the ingestion of a dose of a ketone monoester on CBF and cerebrovascular reactivity to CO2 in young adults.

ELIGIBILITY:
Inclusion Criteria:

* Having a normal blood pressure (≤125/≤85 mmHg)
* Between the ages of 18 and 35

Exclusion Criteria:

* Individuals who are obese (body mass index > 30 kg/m^2)
* Individuals who smoke
* Individuals with respiratory illnesses
* A history of type 2 diabetes, hypoglycemia, or cardiovascular diseases (i.e. heart attack, stroke)
* Individuals currently following a ketogenic diet or taking ketone supplements
* Individuals with a history of concussion(s) with persistent symptoms
* Individuals participating in elite-level physical training (i.e. varsity athletics)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2024-01-19 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Resting cerebral blood flow (CBF) | 90-minutes
  Measured via duplex ultrasound of the internal carotid artery and vertebral artery

SECONDARY OUTCOMES:
Plasma beta-hydroxybutyrate area under the curve | 90-minutes
  Venous blood samples will be obtained via intravenous catheter
Blood pH | 90-minutes
  Venous blood samples will be obtained via intravenous catheter
End-tidal CO2 | 90-minutes
  Breath-by-breath analysis performed via RespirAct (RespirAct, Thornhill Research, Toronto, ON, Canada).
Mean arterial pressure (MAP) | 90-minutes
  Automated blood pressure cuff measurements of brachial artery pressure in mmHg
Cerebrovascular Reactivity of the Internal Carotid and Middle Cerebral Artery as assessed by Duplex Ultrasound and Transcranial Doppler Ultrasound, respectively. | 90-minutes
  Automated gas-blender used to apply sequential gas delivery using an algorithm to target end-tidal CO2 at +3mmHg, +6mmHg, and +9mmHg above baseline, using five-minute step-wise stages. Simultaneously, changes in cerebral blood flow in the internal carotid artery and the middle cerebral artery will be assessed using duplex ultrasound and transcranial Doppler ultrasound, respectively. The final minute of each stage will be analyzed to characterize the slope of cerebrovascular reactivity to CO2 in the internal carotid artery and the middle cerebral artery.
Middle Cerebral Artery Blood Velocity | 90-minutes
  Measured via transcranial Doppler Ultrasound using a 2MHz probe

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy J Walsh, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share individual patient data (de-identified) with researchers upon request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 12 months and ending 36 months following article publication.
Access Criteria: Anyone who wishes to access the data.